CLINICAL TRIAL: NCT04731077
Title: Global, Multicenter, and Prospective Post-Market Clinical Follow-Up Study of the Avenir Complete™ Femoral Stem (Implants and Instrumentation)
Brief Title: Avenir Complete Post-Market Clinical Follow-Up Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMG2020-20H
Record Dates: First submitted 2021-01-28; First posted 2021-01-29 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Osteoarthritis, Hip; Avascular Necrosis of Hip; Avascular Necrosis of the Femoral Head; Post-traumatic; Arthrosis
MeSH Terms: conditions — Osteoarthritis, Hip; Femur Head Necrosis; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Avenir Complete Femoral Stem (Other): All enrolled subjects receive the study implant
  Interventions: Device: Avenir Complete Femoral Stem

INTERVENTIONS:
Device: Avenir Complete Femoral Stem — All enrolled subjects will receive the Avenir Complete Femoral Stem

SUMMARY:
The main objectives of this study are to confirm the long-term safety, performance and clinical benefits the Avenir Complete femoral stem and its instrumentation when used in primary total, hemi, and revision hip arthroplasty.

DETAILED DESCRIPTION:
The main objectives of this study are to confirm the long-term safety, performance and clinical benefits the Avenir Complete™ femoral stem and its instrumentation when used in primary total, hemi, and revision hip arthroplasty:

The primary endpoint is defined by the survival of the implant system at 10 years, which is based on the removal or intended removal of the "study device and determined using Kaplan Meier method. The safety of the system will be assessed by monitoring the frequency and incidence of adverse events. Relation of the events to implant, instrumentation and/or procedure should be specified.

The secondary endpoints are the assessment of performance and clinical benefits by recording patient-reported clinical outcomes measures (PROMs) as well as radiographic outcomes (if available).

ELIGIBILITY:
Inclusion Criteria:

* Patient is at least 20 years old or older and skeletally mature.
* Advanced wear of the joint due to degenerative, post-traumatic or rheumatic diseases;
* Failed previous hip surgery including

  * Joint reconstruction (osteotomy)
  * Arthrodesis
  * Hemi-arthroplasty or total hip replacement (THR)
* Acute traumatic fracture of the femoral head or neck;
* Avascular necrosis of the femoral head.
* Patients capable of understanding the surgeon's explanations and following his instructions, able and willing to participate in the follow-up program and who gave consent to take part in the study;

Exclusion Criteria:

* Acute, chronic, local, or systemic infections;
* Severe muscular, neural, or vascular diseases that endanger the limbs involved;
* Lack of bony structures proximal or distal to the joint, so that good Inclusion criteria
* Patient is at least 20 years old or older and skeletally mature.
* Advanced wear of the joint due to degenerative, post-traumatic or rheumatic diseases;
* Failed previous hip surgery including

  * Joint reconstruction (osteotomy)
  * Arthrodesis
  * Hemi-arthroplasty or total hip replacement (THR)
* Acute traumatic fracture of the femoral head or neck;
* Avascular necrosis of the femoral head.
* Patients capable of understanding the surgeon's explanations and following his instructions, able and willing to participate in the follow-up program and who gave consent to take part in the study;

Exclusion criteria

* Acute, chronic, local, or systemic infections;
* Severe muscular, neural, or vascular diseases that endanger the limbs involved;
* Lack of bony structures proximal or distal to the joint, so that good anchorage of the implant is unlikely or impossible;
* Total or partial absence of the muscular or ligamentous apparatus;
* Any concomitant diseases that can jeopardize the functioning and the success of the implant;
* Allergy to the implanted material, especially to metal (e.g. cobalt, chromium, nickel, etc.);
* Local bone tumors and/or cysts;
* Pregnancy;
* Skeletal immaturity.
* Patients unwilling or unable to give consent, or to comply with the follow-up program;
* Patients who have any condition that would - in the judgement of the Investigator - place him/her at undue risk or
* interfere with the study;
* Any vulnerable subject:

  * a prisoner
  * mentally incompetent or unable to understand what participation in the study entails
  * a known alcohol or drug abuser
  * anticipated to be non-compliant
* Patients with plans to relocate during the study follow-up period;
* Individuals whose willingness to volunteer in a clinical investigation could be unduly influenced by the expectation, whether justified or not, of benefits associated with participation or of retaliatory response from senior members of a hierarchy in case of refusal to participate;

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 275 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2035-06-01 (Estimated); Study Completion 2036-06-01 (Estimated)

PRIMARY OUTCOMES:
Survival of the study device; whether or not it is still implanted in the subject | 10 years
  Survival is classified as removal of the study device for any reason

SECONDARY OUTCOMES:
Incidence of treatment-emergent Adverse Events (safety) | 10 years
  Safety is assessed by monitoring the frequency and incidence of all adverse events, with particular focus on those that may be related to the study device.
Harris Hip Score | 3 years
  Functional outcomes are measured with the Harris Hip Score, including range of motion, pain level, activity levels and patient satisfaction. The score has a maximum of 100 points (best possible outcome) covering pain (1 item, 0-44 points), function (7 items, 0-47 points), absence of deformity (1 item, 4 points), and range of motion (2 items, 5 points).
Patient Quality of Life | 10 years
  This is another self-assessment by means of the EQ-5D-5L (EuroQol) score, which measures the patient's perceived quality of life.
  EQ VAS: Score between 0 and 100 recorded by an individual, 100 being the highest.
  EQ 5D Value: "The value attached to an EQ-5D profile according to a set of weights that reflect, on average, people's preferences about how good or bad the state is. Values are anchored at 1 (full health) and 0 (a state as bad as being dead)" https://euroqol.org/support/terminology/
Radiographic analysis | 10 years
  Postoperative radiographs will be analyzed by the Investigator
Oxford Hip Score | 10 years
  The Oxford Hip Score (OHS) is a joint-specific, patient-reported outcome measure tool designed to assess disability in patients undergoing total hip replacement.
  The score is measured on a scale of 0 to 48 with 48 being the best outcome.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (3):
  - Mississippi Sports Medicine and Orthopaedic Center PLLC, Jackson, Mississippi
  - Heartland Regional Medical Center d.b.a. Mosaic Life Care, Saint Joseph, Missouri
  - Orthopedic & Fracture Clinic, PC, Portland, Oregon
- Copenhagen University Hospital, Hvidovre, Copenhagen, Denmark
- Japan (2):
  - Nissan Tamagawa Hospital, Setagaya-Ku, Tokyo
  - Okayama City Hospital, Okayama
- Ikazia Ziekenhuis, Rotterdam, South Holland, Netherlands
- Sykehuset Innlandet HF, Tynset, Norway
- Sahlgrenska University Hospital - Molndal, Mölndal, Sweden

IPD SHARING:
Plan to Share IPD: No